CLINICAL TRIAL: NCT02607475
Title: Evaluation of Robotic Telesonography for Obstetric and Adult and Pediatric Abdominal Imaging
Brief Title: Evaluation of Robotic Telesonography
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Paul Babyn, Professor, University of Saskatchewan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RT-01
Record Dates: First submitted 2015-11-10; First posted 2015-11-18 (Estimated); Last update posted 2021-10-07 (Actual); Status verified 2021-09

CONDITIONS: Adult Abdominal Imaging; Pediatric Abdominal Imaging; Obstetric Imaging
Keywords: telesonography; ultrasound; robotic telesonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Robotic telesonography compared to conventional sonography (Experimental): All participants will receive two imaging studies: (1) Robotic telesonography using the MELODY Patient System (AdEchoTech) in conjunction with the SonixTablet ultrasound system (BK Ultrasound, formerly Ultrasonix), and (2) conventional sonography using EPIQ 5 (Philips) or LOGIQ E9 (GE Healthcare).
  Interventions: Device: Robotic telesonography (MELODY Patient System, AdEchoTech); Device: Conventional sonography (EPIQ 5, Philips or LOGIQ E9, GE Healthcare)

INTERVENTIONS:
Device: Robotic telesonography (MELODY Patient System, AdEchoTech) — Robotic telesonography using the MELODY Patient System (AdEchoTech) in conjunction with the SonixTablet ultrasound system (BK Ultrasound, formerly Ultrasonix).
Device: Conventional sonography (EPIQ 5, Philips or LOGIQ E9, GE Healthcare) — Conventional sonography using EPIQ 5 (Philips) or LOGIQ E9 (GE Healthcare) ultrasound systems.

SUMMARY:
Robotic telesonography, in which an expert remotely performs sonography in real time, has recently emerged as an opportunity to perform sonography at remote centres. Using a robotic system and an assistant with limited training at the remote site, an expert can manipulate an ultrasound probe and generate images in real-time via an Internet connection. This study aims to demonstrate the feasibility of robotic telesonography for obstetric and adult and pediatric abdominal imaging in a centre with established sonography services which will be used as a comparator to robotic telesonography.

DETAILED DESCRIPTION:
Lack of trained sonographers in remote communities limits access to sonography for many patients. As a result, patients must travel or be transported to secondary and tertiary care centres, which often delays diagnosis and subsequent treatment, creates burdens for patients and their families, and increases healthcare costs. Robotic telesonography, in which an expert remotely performs sonography in real time, has recently emerged as an opportunity to provide sonography regardless of the availability of a skilled operator at the site. Studies primarily originating in Europe have demonstrated robotic telesonography in abdominal, pelvic, obstetric, and cardiologic applications in adults. However, the full potential of robotic telesonography across many imaging applications has yet to be explored, and robotic telesonography has not yet been trialed in Canada. This study aims to demonstrate the feasibility of robotic telesonography in a centre with established sonography services which will be used as a comparator to robotic telesonography. Approximately 30 patients will be recruited for each substudy (obstetric, adult abdominal, and pediatric abdominal). All patients will receive both conventional and robotic scans in a crossover design. The sonographer performing the scan will be asked to complete a data collection form which will collect information about duration of the exam and any challenges encountered. Following the completion of both scans, the patient-site assistant will provide a questionnaire to the patient (or for children, a parent/guardian of the patient) regarding his/her experience with the system. A physician will review images generated using either the robotic telesonography or conventional sonography systems and report findings on a standardized reporting form.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to have an abdominal study or second trimester ultrasound study at Royal University Hospital or Saskatoon Medical Imaging.
* Pediatric abdominal substudy: male and female patients 5 years of age or older and less than 18 years of age
* Adult abdominal substudy: male and female patients 18 years of age and older
* Obstetrics substudy: second trimester patients 18 years of age and older

Exclusion Criteria:

* Patients who do not meet the inclusion criteria above
* Patients who are in distress prior to or during the exam

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2015-11; Primary Completion 2022-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance of robotic telesonography, expressed as the concordance of measurements and concordance of findings visualized with robotic telesonography using conventional sonography as a reference standard. | Research images will be interpreted within 8 weeks

SECONDARY OUTCOMES:
Duration of robotic telesonography exams relative to conventional sonography | 1 day
Acceptability of the robotic telesonography experience to patients measured using Likert items | 1 day
Acceptability of the robotic telesonography system to remote users (sonographers) and patient-site assistants measured using Likert items | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Paul S. Babyn, MDCM, FRCPC, Principal Investigator — University of Saskatchewan
Locations (3):
- Canada (3):
  - Saskatoon Medical Imaging, Saskatoon, Saskatchewan
  - Royal University Hospital, Saskatoon, Saskatchewan
  - The Ultrasound Centre, Saskatoon, Saskatchewan